CLINICAL TRIAL: NCT06765863
Title: Low Birthweight and Preterm Infant Feeding Trial and Supportive Care Package (LIFT-UP): Randomized Controlled Trial of In-facility Fortification of Human Milk in India
Brief Title: LIFT-UP: Randomized Controlled Trial of Fortification of Human Milk
Acronym: LIFT-UP RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Boston Children's Hospital (Other); Brigham and Women's Hospital (Other); Emory University (Other); Muhimbili University of Health and Allied Sciences (Other); Jawaharlal Nehru Medical College (Other); PATH (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, Katherine Semrau, Deputy Director, Ariadne Labs & Director, BetterBirth Program; Associate Professor, HSPH, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB23-0304
Record Dates: First submitted 2024-12-26; First posted 2025-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Very Preterm Infant; Very Low Birthweight
Keywords: very preterm; very low birthweight; fortification; human milk

STUDY DESIGN:
Intervention Model Description: Mother-infant dyads will be individually randomized 1:1 to the intervention or comparison arm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants (i.e. mother-infant dyads) will not be blinded and will know if the fortification is being provided to the infant as it will be mixed with human milk [MOM or PHDM] in the intervention arm. Clinical research staff will not be blinded as they are preparing and providing the intervention and control feeding assignments. Data collectors and the analysis team will be blinded to study arm assignments to reduce bias in data collection and analysis. These individuals (data collectors and analysis team) will be independent from the clinical study staff who are providing the intervention or control. For data analysis, groups will be labeled with a letter (A vs B) to conceal allocation assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine fortification of human milk with human milk fortifier using a standardized clinical protocol (Experimental): Enrolled participants in the intervention arm will be exposed to:
  * Provision of guideline-driven standard of care specifically for VPT/ VLBW babies
  * Encouragement to express breast milk with breast pumps
  * Adherence to a clinical guideline including targets for initiation and advancement of breast milk feeding for VPT/ VLBW babies based on birthweight
  * Fortification of human milk with HMF
  * Adherence to standardized stopping criteria (i.e., stopping adherence to clinical feeding guideline AND stopping routine fortification of human milk)
  Interventions: Dietary Supplement: Human Milk Fortifier; Other: Volume targets
- No routine fortification of human milk using a standardized clinical protocol (Active Comparator): Participants in the control group will have the same exposures as the participants in the intervention group EXCEPT for the human milk consumed will not be fortified with HMF.
  * Provision of guideline-driven standard of care specifically for VPT/ VLBW babies
  * Encouragement to express with breast pumps
  * Adherence to a clinical guideline including targets for initiation and advancement of breast milk feeding for VPT/ VLBW babies based on birthweight
  * Adherence to standardized stopping criteria (i.e., stopping adherence to clinical feeding guideline)
  Interventions: Other: Volume targets

INTERVENTIONS:
Dietary Supplement: Human Milk Fortifier — Human milk fortifier added to expressed human milk (mother's own milk or pasteurized donor human milk) per feed per manufacturer's instructions for a minimum of 21 days (in-facility provision only)
  * Clinical feeding guideline including targets for initiation and advancement of breast milk feeding
  * Provision of guideline-driven standard of care [facility-based lactation support/feeding counseling + KMC + WASH package (referred to as facility-based FSP+) and breast pumps]
  Other Names: Volume targets; Guideline-driven standard of care
  Arms: Routine fortification of human milk with human milk fortifier using a standardized clinical protocol
Other: Volume targets — * Clinical feeding guideline including targets for initiation and advancement of breast milk feeding
  * Provision of guideline-driven standard of care [facility-based lactation support/feeding counseling + KMC + WASH package (referred to as facility-based FSP+) and breast pumps]
  Other Names: Guideline driven standard of care

SUMMARY:
The goal of the LIFT-UP randomized controlled trial is to evaluate the efficacy of feeding routinely and fortified human milk using a standardized clinical protocol to very low birthweight (VLBW) or very preterm (VPT) infants in the NICU compared to not feeding routinely fortified human milk using the standardized clinical protocol.

The primary research question is: Will VLBW or VPT infants in the NICU who are fed fortified human milk using a standardized feeding protocol have better growth outcomes by facility discharge and at 3 months of age, less illness by discharge, and decreased mortality by discharge and at one month compared to those who are not routinely fed fortified human milk using the same feeding protocol?

DETAILED DESCRIPTION:
AIM: To improve feeding and growth outcomes among very low birthweight (LBW; ≤1.5kg) or very preterm (≤32 weeks gestational age) infants admitted to neonatal intensive care units (NICU) in India through fortification of human milk.

OBJECTIVE: To evaluate (via individually randomized controlled study) the efficacy of feeding routinely and fortified human milk using a standardized clinical protocol to very LBW or very preterm infants in the NICU compared to not feeding routinely fortified human milk using the standardized clinical protocol.

STUDY DESIGN This study is a multi-site individually randomized prospective trial among VLBW or VPT infants admitted to the NICU in study facilities who consume human milk and meet eligibility criteria (along with their mothers).

SCREENING AND ENROLLMENT All infants admitted to the NICU and their mothers will be screened for study eligibility. Screening will be performed within 24 hours of birth for inborn infants and within 48 hours of birth for outborn infants. Eligible dyads with the intention to feed human milk [mother's own milk (MOM) or pasteurized donor human milk (PDHM)] whose mothers provide consent will be enrolled into the study.

Once the mother-infant dyad is enrolled and prior to randomization, they will:

Receive the guideline-driven standard of care and be provided access to breast pumps to help initiate and advance breast milk feeding. The guideline-driven standard of care includes facility-based lactation support/feeding counseling + KMC + WASH components designed specifically for small vulnerable newborns and was developed as part of a different study protocol (see NCT06390943).

Adhere to a clinical guideline including targets for initiating and advancing breast milk feeding. Initially, this clinical guideline will help infants achieve breast milk volume intake of at least 60 mL/kg/day, the primary criterion for randomization. After randomization, the clinical guideline will continue to support advancing human milk feeding for all infants advance to 180 mL/kg/day.

RANDOMIZATION Once an infant consumes at least 60 mL/kg/day of breast milk, enrolled dyads will be assessed for eligibility for randomization. Eligible dyads will be randomized individually in a 1:1 ratio to either the intervention or comparison arm. Randomization sequences will be previously generated by the study statistician. If an infant does not consume at least 60 mL/kg/day of breastmilk by day 10 of chronological age, the mother-infant dyad will be administratively withdrawn from the study.

DELIVERY OF INTERVENTION Mothers of infants randomized to the intervention arm will express their breast milk into a standardized measurement cup (or PDHM can be used). Clinical research staff will mix human milk fortifier (HMF) in human milk (either MOM or PDHM, if available) per manufacturer specifications per feed for a minimum of 21 days.

Dyads in both arms will continue to receive the guideline-driven standard of care, access to breast pumps, and follow the volume target and trajectory protocol until they meet stopping criteria. Data will be collected every 24 hours, including a log at every feed, regardless of study arm assignment.

If an infant in either arm does not meet protocolized minimum volume targets or trajectories AND that infant meets weight-based safety net criteria, clinicians will intervene per judgment aligned with national and local protocols.

The intervention will not be continued once the infant meets stopping criteria with the goal of the infant having fully transitioned to exclusive breast milk feeding by then.

STOPPING CRITERIA After the minimum duration of 21 days post-randomization, hospitalized infants should continue to receive volume targeted feeding with or without HMF for as long as they receive expressed breast milk. Once infants transition to full, direct breastfeeding in preparation for discharge or are being discharged per clinician discretion, they will stop adhering to the volume targets and infants in the intervention group will stop receiving fortified human milk.

DISCHARGE FROM FACILITY TO HOME After stopping criteria are met, routine clinical care around infant feeding will be provided. Infants can be discharged home when deemed clinically appropriate per facility protocols and clinician judgment. The guideline-driven standard of care will encourage all mothers to exclusively breastfeed their infants prior to discharge and to continue doing so after discharge.

POST-DISCHARGE FACILITY VISITS All dyads will be followed up at 2 weeks of age, 4 weeks of age, and 3 months of chronological age.

ELIGIBILITY:
Inclusion Criteria:

* Very LBW (≤1.5kg)* or very preterm (≤32 weeks) infants admitted to NICU at study facility within 24 hours of birth for in-born infants and up to 48 hours for out-born**
* Mother and infant alive during screening
* Mother age 18+ years
* Lives within catchment areas of the facility
* Mother intends to stay in catchment area of the study facility for at least 3 months
* At randomization: Infant receiving at least 60 mL/kg/day of human milk***

Exclusion Criteria:

* Lives outside the defined catchment area
* Congenital abnormalities or acquired conditions that interfere with feeding or placement of nasogastric/orogastric tube [cleft lip/palate, toxoplasmosis, other agents, rubella, cytomegalovirus, and herpes (TORCH), Trisomy 21, congenital cardiac defect, neural tube defect, gastrointestinal tract anomalies, hydrocephalus, NEC]
* Severe birth asphyxia
* Critically ill (i.e. not on enteral feeds)
* Unknown date of birth and unknown gestational age

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 776 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Length-for-age Z score (LAZ) | 3 Months
  Mean LAZ (SD, range) measured at birth, 2 weeks, 4 weeks and 3 months of age

SECONDARY OUTCOMES:
Length of Stay | From date of randomization until the date of facility discharge or date of death from any cause, whichever came first, assessed up to 3 months of age.
  Mean (SD) number of days admitted in the study facility from randomization to facility discharge
Feeding intolerance | From randomization to facility discharge, assessed up to 3 months of age
  % infants identified with feeding intolerance
Weight growth velocity | From randomization to facility discharge, assessed up to 3 months of age
  % infants attaining 15 g/kg/day
Length gain | From randomization to facility discharge, assessed up to 3 months of age.
  Mean (SD) change in length (mm/week)
Head circumference gain | From randomization to facility discharge, assessed up to 3 months of age
  Mean (SD) change in head circumference (mm per week)
Necrotizing enterocolitis (NEC) | From randomization to facility discharge, assessed up to 3 months of age.
  % infants diagnosed with NEC
Sepsis/possible serious bacterial infection (PSBI) | From randomization to facility discharge, assessed up to 3 months of age
  % diagnosed with sepsis or possible serious bacterial infection (PSBI)
Infant mortality | From randomization to 3 months of age
  % infants died
Birthweight regain | 2 weeks of age
  % infants who regain birthweight by 2 weeks of age
Mean weight growth velocity (4 weeks) | From randomization to 4 weeks of age
  Mean (SD) change in weight (growth) at 4 weeks of age
Neonatal mortality (4 weeks) | From randomization to 4 weeks of age
  % of neonates who died up to 4 weeks of age
Sepsis/possible serious bacterial infection (PSBI, 4 weeks) | From randomization to 4 weeks of age
  % of infants diagnosed with sepsis/PSBI up to 4 weeks of age
Mean weight growth velocity | From randomization to facility discharge, assessed up to 3 months of age.
  Mean change in infant weight (growth) calculated in grams/kilogram/day (g/kg/day)
Weight-for-age Z score (WAZ) | 3 months of age
  Mean (SD) WAZ at 3 months of age
Weight-for-length Z score (WLZ) | 3 months of age
  Mean (SD) weight-for-length Z score (WLZ) at 3 months of age
Head circumference-for-age Z score (HcAZ) | 3 months of age
  Mean (SD) HcAZ
Change in WAZ | From randomization to 3 months of age
  Change in WAZ from randomization to 3 months of age
Change in LAZ | From randomization to 3 months of age
  Change in LAZ from randomization to 3 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Semrau, PhD, MPH, Principal Investigator — Ariadne Labs | Harvard TH Chan School of Public Health and Brigham and Womens Hospital
Locations (4):
- India (4):
  - Ballari Medical College and Research Centre, Ballary, Karnataka
  - KLES Dr Prabhakar Kore Hospital & Medical Research Center, Belagavi, Karnataka
  - JJM Medical College, Davangere, Karnataka
  - Niloufer Hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be released after the close of the project in a data sharing repository, such as Harvard Dataverse or similar, in a format readable by analytics tools. Harvard Dataverse is an online data repository where you can share, preserve, cite, explore, and analyze research data. Datasets and data dictionaries will be provided in compliance with the ethical review board requirements. As part of the Harvard Dataverse system, registration to download datasets is required. External partners (those not involved in the study) must provide their contact information and describe their intention of data use.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Study data will be available after study completion, expected in mid-2027.
Access Criteria: Data will be available on Harvard Dataverse and users will register for access stating their intent to use the data.